CLINICAL TRIAL: NCT05763875
Title: A Double-blind, Randomized, Placebo- and Active-Comparator Controlled Study to Evaluate the Efficacy of Inclisiran as Monotherapy in Patients With Primary Hypercholesterolemia Not Receiving Lipid-Lowering Therapy (VictORION-Mono)
Brief Title: Efficacy and Safety of Inclisiran as Monotherapy in Patients With Primary Hypercholesterolemia Not Receiving Lipid-lowering Therapy.
Acronym: V-Mono
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CKJX839D12304
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Hypercholesterolemia
Keywords: inclisiran; ezetimibe; LDL-C; monotherapy; primary hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — ALN-PCS; Ezetimibe

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized, double-blind, placebo- and active comparator-controlled, parallel groups
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sponsor Personnel participating in the study conduct were also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Inclisiran (Experimental): Inclisiran s.c and Placebo p.o
  Interventions: Drug: Inclisiran; Drug: Matching Placebo for Ezetimibe
- Ezetimibe (Active Comparator): Placebo s.c. and Ezetimibe p.o.
  Interventions: Drug: Ezetimibe; Drug: Matching Placebo for Inclisiran
- Placebo (Placebo Comparator): Placebo s.c. and Placebo p.o.
  Interventions: Drug: Matching Placebo for Inclisiran; Drug: Matching Placebo for Ezetimibe

INTERVENTIONS:
Drug: Inclisiran — 284 mg (equivalent to 300 mg inclisiran sodium) subcutaneous injection given on Day 1 and Day 90
  Other Names: KJX839
  Arms: Inclisiran
Drug: Ezetimibe — 10 mg over-encapsulated tablet taken once a day from Day 1 through Day 149
  Other Names: Sandoz ezetimibe
  Arms: Ezetimibe
Drug: Matching Placebo for Inclisiran — 0mg placebo injection solution for subcutaneous injection on Day 1 and Day 90
  Other Names: Placebo s.c.
  Arms: Ezetimibe; Placebo
Drug: Matching Placebo for Ezetimibe — 0mg over-encapsulated placebo tablet taken once a day from Day 1 through Day 149
  Other Names: Placebo p.o.
  Arms: Inclisiran; Placebo

SUMMARY:
CKJX839D12304 was a research study to determine if the study treatment, called inclisiran, in comparison to placebo and ezetimibe effectively reduces Low-Density Lipoprotein Cholesterol (LDL-C) as measured by percentage change from baseline to Day 150. This study was conducted in eligible participants with primary hypercholesterolemia not receiving any lipid-lowering therapy (LLT), with a 10-year Atherosclerotic Cardiovascular Disease (ASCVD) risk of less than 7.5%.

DETAILED DESCRIPTION:
This study was a randomized, double-blind, placebo- and active comparator-controlled, multicenter study in 350 adult participants with primary hypercholesterolemia not receiving any LLT with a 10-year ASCVD risk score of less than 7.5%. This study evaluated the efficacy and safety of inclisiran sodium 300 mg, administered as a monotherapy in comparison to ezetimibe and placebo.

The study consisted of:

* a screening period of up to 14 days;
* a double-blind treatment period of 150+/- 5 days during which participants were randomly assigned to either the inclisiran arm, the ezetimibe arm or the placebo arm in a 2:1:1 ratio; and
* a safety follow-up / End of Study visit conducted 30+5 days after the Day 150 visit.

The overall study duration was approximately 190 days.

ELIGIBILITY:
Inclusion Criteria at screening:

* informed consent signed prior to participation in study
* fasting LDL-C of >= 100 mg/dL but < 190 mg/dL
* fasting triglycerides <= 400 mg/dL
* 10-year ASCVD risk score < 7.5%
* not on any lipid-lowering therapy within 90 days of screening

Key Exclusion Criteria:

* history of ASCVD
* diabetes mellitus or fasting plasma glucose of >= 7.0 mmol/L or HbA1c >= 6.5%
* secondary hypercholesterolemia, e.g. hypothyroidism (TSH above upper limit of normal)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (41):
- United States (22):
  - Parkway Medical Center, Birmingham, Alabama
  - SEC Clinical Research, Dothan, Alabama
  - Hillcrest Medical Research, DeLand, Florida
  - ClinCloud, Maitland, Florida
  - Alma Clinical Research Inc, Miami, Florida
  - Inpatient Research Clinical LLC, Miami Lakes, Florida
  - Harmony Clinical Research, North Miami Beach, Florida
  - Fam Medical Specialists Of Fl Plc, Plant City, Florida
  - Cozy Research LLC, Zephyrhills, Florida
  - Koch Family Medicine, Morton, Illinois
  - Grace Research LLC, Bossier City, Louisiana
  - Grace Research Llc, Shreveport, Louisiana
  - Southern Clin Research Clinic, Zachary, Louisiana
  - Prime Global Research Inc, The Bronx, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - WellNow Urgent Care and Research, Huber Heights, Ohio
  - Conrad Clinical Research, Edmond, Oklahoma
  - Compass Point Research, Nashville, Tennessee
  - Mt Olympus Medical Research, Sugar Land, Texas
  - Dominion Medical Associates, Richmond, Virginia
  - Spaulding Clinical Research, West Bend, Wisconsin
- Colombia (4):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Floridablanca, Santander Department
  - Novartis Investigative Site, Manizales
  - Novartis Investigative Site, San Gil
- Germany (9):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Löhne, North Rhine-Westphalia
  - Novartis Investigative Site, Jerichow, Saxony-Anhalt
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Gladbeck
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Papenburg
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Pécs
- Mexico (4):
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Mérida, Yucatán
  - Novartis Investigative Site, Culiacan Sinaloa
  - Novartis Investigative Site, Querétaro

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Taub PR, Gutierrez A, Wewers D, Garcia Cantu E, Cao H, Deck C, Lesogor A, Ott D, Mena-Madrazo J, Zang X, Wright RS. Safety and Lipid-Lowering Efficacy of Inclisiran Monotherapy in Patients Without ASCVD: The VICTORION-Mono Randomized Clinical Trial. J Am Coll Cardiol. 2025 Jul 22;86(3):196-208. doi: 10.1016/j.jacc.2025.04.049. Epub 2025 May 5. PMID 40392667
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2658

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 42 investigative sites in 5 countries
Pre-assignment Details: There was a 14 day screening period
Period: Overall Study
Arm/Group | Inclisiran | Ezetimibe | Placebo
Started | 174 | 89 | 87
Completed | 164 | 86 | 84
Not Completed | 10 | 3 | 3
Not completed — Subject decision | 5 | 2 | 1
Not completed — Lost to Follow-up | 4 | 1 | 2
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inclisiran | Ezetimibe | Placebo | Total
Number analyzed (Participants) | 174 | 89 | 87 | 350
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 168 | 86 | 83 | 337
  >=65 years | 6 | 3 | 4 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (11.74) | 46.3 (10.90) | 46.7 (11.55) | 46.1 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 56 | 59 | 219
  Male | 70 | 33 | 28 | 131
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 10 | 9 | 29
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 20 | 7 | 10 | 37
  White | 140 | 71 | 67 | 278
  More than one race | 4 | 0 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline Low-Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 135.8 (27.01) | 134.4 (25.82) | 135.4 (28.69) | 135.4 (27.07)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Low-density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 150
Description: Percentage change in LDL-C from Baseline (day 1) to Day 150, Inclisiran arm versus Ezetimibe and placebo.
  There were two estimands of interest in comparing efficacy of inclisiran as monotherapy against that of placebo or ezetimibe that differ on the treatment of interest used for each and the management of intercurrent events as follows:
  * Monotherapy Estimand: Inclisiran as monotherapy compared to the use of comparator. This estimand uses a hypothetical strategy where participants who permanently discontinued treatment, died or used other LLTs were handled in a hypothetical scenario of what would have happened if the intercurrent event did not happen.
  * Treatment-policy Estimand: Inclisiran as monotherapy compared to the use of comparator with or without other lipid lowering therapies (LLTs) added. This estimand ignored the use of other LLTs and treatment discontinuation. Deaths (if any) were handled as an unfavorable outcome using a composite variable strategy.
Time Frame: Baseline, Day 150
Population: Full Analysis Set, all randomized participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change from baseline
Arm/Group | Inclisiran | Ezetimibe | Placebo
Number analyzed (Participants) | 174 | 89 | 87
Percentage change from baseline
  LS Mean (Treatment Policy estimand) | -46.54 [-50.20 to -42.88] | -11.17 [-15.34 to -7.00] | 1.37 [-3.07 to 5.80]
  LS Mean (Monotherapy estimand) | -49.37 [-52.76 to -45.97] | -11.92 [-15.87 to -7.98] | -1.53 [-2.97 to 6.03]
Statistical Analysis 1: Comparison: Inclisiran vs Ezetimibe; Treatment Policy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -35.37, 95% CI 2-sided [-40.88 to -29.86]
Statistical Analysis 2: Comparison: Inclisiran vs Placebo; Treatment Policy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -47.91, 95% CI 2-sided [-53.62 to -42.20]
Statistical Analysis 3: Comparison: Inclisiran vs Ezetimibe; Monotherapy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -37.44, 95% CI 2-sided [-42.63 to -32.26]
Statistical Analysis 4: Comparison: Inclisiran vs Placebo; Monotherapy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -50.90, 95% CI 2-sided [-56.51 to -45.28]

2. Secondary Outcome: Absolute Change in LDL-C From Baseline to Day 150
Description: Absolute change in LDL-C from Baseline (Day 1) to Day 150, Inclisiran arm versus Ezetimibe and placebo.
  There were two estimands of interest in comparing efficacy of inclisiran as monotherapy against that of placebo or ezetimibe that differ on the treatment of interest used for each and the management of intercurrent events as follows:
  * Monotherapy Estimand: Inclisiran as monotherapy compared to the use of comparator. This estimand uses a hypothetical strategy where participants who permanently discontinued treatment, died or used other LLTs were handled in a hypothetical scenario of what would have happened if the intercurrent event did not happen.
  * Treatment-policy Estimand: Inclisiran as monotherapy compared to the use of comparator with or without other lipid lowering therapies (LLTs) added. This estimand ignored the use of other LLTs and treatment discontinuation. Deaths (if any) were handled as an unfavorable outcome using a composite variable strategy.
Time Frame: Baseline, Day 150
Population: Full Analysis Set, all randomized participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran | Ezetimibe | Placebo
Number analyzed (Participants) | 174 | 89 | 87
mg/dL
  LS Mean (Treatment Policy estimand) | -64.86 [-69.27 to -60.46] | -17.55 [-22.53 to -12.57] | -1.29 [-6.40 to 3.82]
  LS Mean (Monotherapy estimand) | -68.57 [-72.59 to -64.56] | -18.52 [-23.16 to -13.89] | -1.07 [-6.32 to 4.19]
Statistical Analysis 1: Comparison: Inclisiran vs Ezetimibe; Treatment Policy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -47.37, 95% CI 2-sided [-53.91 to -40.72]
Statistical Analysis 2: Comparison: Inclisiran vs Placebo; Treatment Policy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -63.57, 95% CI 2-sided [-70.28 to -56.87]
Statistical Analysis 3: Comparison: Inclisiran vs Ezetimibe; Monotherapy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -50.05, 95% CI 2-sided [-56.16 to -43.94]
Statistical Analysis 4: Comparison: Inclisiran vs Placebo; Monotherapy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -67.51, 95% CI 2-sided [-74.09 to -60.92]

3. Secondary Outcome: Percentage Change in Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) From Baseline to Day 150
Description: Percentage change in PCSK9 from Baseline (Day 1) to Day 150 , Inclisiran arm versus Ezetimibe and placebo.
  There were two estimands of interest in comparing efficacy of inclisiran as monotherapy against that of placebo or ezetimibe that differ on the treatment of interest used for each and the management of intercurrent events as follows:
  * Monotherapy Estimand: Inclisiran as monotherapy compared to the use of comparator. This estimand uses a hypothetical strategy where participants who permanently discontinued treatment, died or used other LLTs were handled in a hypothetical scenario of what would have happened if the intercurrent event did not happen.
  * Treatment-policy Estimand: Inclisiran as monotherapy compared to the use of comparator with or without other lipid lowering therapies (LLTs) added. This estimand ignored the use of other LLTs and treatment discontinuation. Deaths (if any) were handled as an unfavorable outcome using a composite variable strategy.
Time Frame: Baseline, Day 150
Population: Full Analysis Set, all randomized participants with a valid assessment for the outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change from baseline
Arm/Group | Inclisiran | Ezetimibe | Placebo
Number analyzed (Participants) | 172 | 89 | 87
Percentage change from baseline
  LS Mean (Treatment Policy estimand): number analyzed (Participants) | 172 | 89 | 85
  LS Mean (Treatment Policy estimand) | -67.12 [-73.21 to -61.03] | 6.04 [-0.10 to 12.18] | 7.82 [0.35 to 15.29]
  LS Mean (Monotherapy estimand): number analyzed (Participants) | 172 | 89 | 85
  LS Mean (Monotherapy estimand) | -71.31 [-76.73 to -65.89] | 5.56 [-0.67 to 11.79] | 8.16 [0.59 to 15.74]
Statistical Analysis 1: Comparison: Inclisiran vs Ezetimibe; Treatment Policy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -73.16, 95% CI 2-sided [-81.76 to -64.56]
Statistical Analysis 2: Comparison: Inclisiran vs Placebo; Treatment Policy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -74.94, 95% CI 2-sided [-84.51 to -65.37]
Statistical Analysis 3: Comparison: Inclisiran vs Ezetimibe; Monotherapy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -76.87, 95% CI 2-sided [-85.12 to -68.62]
Statistical Analysis 4: Comparison: Inclisiran vs Placebo; Monotherapy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -79.47, 95% CI 2-sided [-88.77 to -70.17]

4. Secondary Outcome: Percentage Change in Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) From Baseline to Day 150
Description: Percentage change in non-HDL-C from Baseline (Day 1) to Day 150, Inclisiran arm versus Ezetimibe and placebo.
  There were two estimands of interest in comparing efficacy of inclisiran as monotherapy against that of placebo or ezetimibe that differ on the treatment of interest used for each and the management of intercurrent events as follows:
  * Monotherapy Estimand: Inclisiran as monotherapy compared to the use of comparator. This estimand uses a hypothetical strategy where participants who permanently discontinued treatment, died or used other LLTs were handled in a hypothetical scenario of what would have happened if the intercurrent event did not happen.
  * Treatment-policy Estimand: Inclisiran as monotherapy compared to the use of comparator with or without other lipid lowering therapies (LLTs) added. This estimand ignored the use of other LLTs and treatment discontinuation. Deaths (if any) were handled as an unfavorable outcome using a composite variable strategy.
Time Frame: Baseline, Day 150
Population: Full Analysis Set, all randomized participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change from baseline
Arm/Group | Inclisiran | Ezetimibe | Placebo
Number analyzed (Participants) | 174 | 89 | 87
Percentage change from baseline
  LS Mean (Treatment Policy estimand) | -40.45 [-43.50 to -37.40] | -9.97 [-13.34 to -6.61] | 1.88 [-2.75 to 6.50]
  LS Mean (Monotherapy estimand) | -42.82 [-45.62 to -40.02] | -10.84 [-13.84 to -7.84] | 2.04 [-2.63 to 6.71]
Statistical Analysis 1: Comparison: Inclisiran vs Ezetimibe; Treatment Policy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -30.48, 95% CI 2-sided [-34.98 to -25.98]
Statistical Analysis 2: Comparison: Inclisiran vs Placebo; Treatment Policy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -42.32, 95% CI 2-sided [-47.83 to -36.82]
Statistical Analysis 3: Comparison: Inclisiran vs Ezetimibe; Monotherapy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -31.98, 95% CI 2-sided [-36.07 to -27.89]
Statistical Analysis 4: Comparison: Inclisiran vs Placebo; Monotherapy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -44.86, 95% CI 2-sided [-50.28 to -39.44]

5. Secondary Outcome: Percentage Change in Total Cholesterol (TC)/HDL-C Ratio From Baseline to Day 150
Description: Percentage change in total cholesterol/HDL-C ratio from Baseline (Day1) to Day 150, Inclisiran arm versus Ezetimibe and placebo.
  There were two estimands of interest in comparing efficacy of inclisiran as monotherapy against that of placebo or ezetimibe that differ on the treatment of interest used for each and the management of intercurrent events as follows:
  * Monotherapy Estimand: Inclisiran as monotherapy compared to the use of comparator. This estimand uses a hypothetical strategy where participants who permanently discontinued treatment, died or used other LLTs were handled in a hypothetical scenario of what would have happened if the intercurrent event did not happen.
  * Treatment-policy Estimand: Inclisiran as monotherapy compared to the use of comparator with or without other lipid lowering therapies (LLTs) added. This estimand ignored the use of other LLTs and treatment discontinuation. Deaths (if any) were handled as an unfavorable outcome using a composite variable strate
Time Frame: Baseline, Day 150
Population: Full Analysis Set, all randomized participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change from baseline
Arm/Group | Inclisiran | Ezetimibe | Placebo
Number analyzed (Participants) | 174 | 89 | 87
Percentage change from baseline
  LS Mean (Treatment Policy estimand) | -31.54 [-35.43 to -27.65] | -6.70 [-10.61 to -2.78] | 2.31 [-4.05 to 8.68]
  LS Mean (Monotherapy estimand) | -33.56 [-37.32 to -29.79] | -6.98 [-10.99 to -2.97] | 2.51 [-3.90 to 8.91]
Statistical Analysis 1: Comparison: Inclisiran vs Ezetimibe; Treatment Policy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -24.84, 95% CI 2-sided [-30.32 to -19.36]
Statistical Analysis 2: Comparison: Inclisiran vs Placebo; Treatment Policy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -33.85, 95% CI 2-sided [-41.27 to -26.44]
Statistical Analysis 3: Comparison: Inclisiran vs Ezetimibe; Monotherapy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -26.58, 95% CI 2-sided [-32.07 to -21.09]
Statistical Analysis 4: Comparison: Inclisiran vs Placebo; Monotherapy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -36.06, 95% CI 2-sided [-43.46 to -28.67]

6. Secondary Outcome: Percentage Change in Apolipoprotein B (Apo B) From Baseline to Day 150
Description: Percentage change in Apo B from Baseline (Day 1) to Day 150, Inclisiran arm versus Ezetimibe and placebo.
  There were two estimands of interest in comparing efficacy of inclisiran as monotherapy against that of placebo or ezetimibe that differ on the treatment of interest used for each and the management of intercurrent events as follows:
  * Monotherapy Estimand: Inclisiran as monotherapy compared to the use of comparator. This estimand uses a hypothetical strategy where participants who permanently discontinued treatment, died or used other LLTs were handled in a hypothetical scenario of what would have happened if the intercurrent event did not happen.
  * Treatment-policy Estimand: Inclisiran as monotherapy compared to the use of comparator with or without other lipid lowering therapies (LLTs) added. This estimand ignored the use of other LLTs and treatment discontinuation. Deaths (if any) were handled as an unfavorable outcome using a composite variable strategy.
Time Frame: Baseline, Day 150
Population: Full Analysis Set, all randomized participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change from baseline
Arm/Group | Inclisiran | Ezetimibe | Placebo
Number analyzed (Participants) | 174 | 89 | 87
Percentage change from baseline
  LS Mean (Treatment Policy estimand) | -37.39 [-40.25 to -34.54] | -8.41 [-11.71 to -5.12] | -0.73 [-4.18 to 2.72]
  LS Mean (Monotherapy estimand) | -39.36 [-42.00 to -36.72] | -9.20 [-12.13 to -6.28] | -0.58 [-4.07 to 2.90]
Statistical Analysis 1: Comparison: Inclisiran vs Ezetimibe; Treatment Policy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -28.98, 95% CI 2-sided [-33.30 to -24.65]
Statistical Analysis 2: Comparison: Inclisiran vs Placebo; Treatment Policy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -36.66, 95% CI 2-sided [-41.10 to -32.22]
Statistical Analysis 3: Comparison: Inclisiran vs Ezetimibe; Monotherapy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -30.16, 95% CI 2-sided [-34.08 to -26.23]
Statistical Analysis 4: Comparison: Inclisiran vs Placebo; Monotherapy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -38.78, 95% CI 2-sided [-43.12 to -34.43]

7. Secondary Outcome: Percentage Change in Apo B/Apo A-1 Ratio From Baseline to Day 150
Description: Percentage change in Apo B/Apo A-1 ratio from baseline (Day 1) to Day 150, Inclisiran arm versus Ezetimibe and placebo.
  There were two estimands of interest in comparing efficacy of inclisiran as monotherapy against that of placebo or ezetimibe that differ on the treatment of interest used for each and the management of intercurrent events as follows:
  * Monotherapy Estimand: Inclisiran as monotherapy compared to the use of comparator. This estimand uses a hypothetical strategy where participants who permanently discontinued treatment, died or used other LLTs were handled in a hypothetical scenario of what would have happened if the intercurrent event did not happen.
  * Treatment-policy Estimand: Inclisiran as monotherapy compared to the use of comparator with or without other lipid lowering therapies (LLTs) added. This estimand ignored the use of other LLTs and treatment discontinuation. Deaths (if any) were handled as an unfavorable outcome using a composite variable strategy.
Time Frame: Baseline, Day 150
Population: Full Analysis Set, all randomized participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change from baseline
Arm/Group | Inclisiran | Ezetimibe | Placebo
Number analyzed (Participants) | 174 | 89 | 87
Percentage change from baseline
  LS Mean (Treatment Policy estimand) | -37.79 [-43.03 to -32.55] | -7.55 [-11.74 to -3.36] | -2.65 [-5.69 to 0.39]
  LS Mean (Monotherapy estimand) | -40.03 [-45.25 to -34.82] | -7.69 [-12.00 to -3.37] | -2.65 [-5.81 to 0.50]
Statistical Analysis 1: Comparison: Inclisiran vs Ezetimibe; Treatment Policy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -30.24, 95% CI 2-sided [-36.92 to -23.57]
Statistical Analysis 2: Comparison: Inclisiran vs Placebo; Treatment Policy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -35.15, 95% CI 2-sided [-41.18 to -29.12]
Statistical Analysis 3: Comparison: Inclisiran vs Ezetimibe; Monotherapy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -32.34, 95% CI 2-sided [-39.10 to -25.59]
Statistical Analysis 4: Comparison: Inclisiran vs Placebo; Monotherapy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -37.38, 95% CI 2-sided [-43.44 to -31.31]

8. Secondary Outcome: Change in Lipoprotein (a) [Lp(a)] From Baseline to Day 150
Description: Day 150 / Baseline ratio in Lp(a) in Inclisiran arm versus Ezetimibe and placebo.
  There were two estimands of interest in comparing efficacy of inclisiran as monotherapy against that of placebo or ezetimibe that differ on the treatment of interest used for each and the management of intercurrent events as follows:
  * Monotherapy Estimand: Inclisiran as monotherapy compared to the use of comparator. This estimand uses a hypothetical strategy where participants who permanently discontinued treatment, died or used other LLTs were handled in a hypothetical scenario of what would have happened if the intercurrent event did not happen.
  * Treatment-policy Estimand: Inclisiran as monotherapy compared to the use of comparator with or without other lipid lowering therapies (LLTs) added. This estimand ignored the use of other LLTs and treatment discontinuation. Deaths (if any) were handled as an unfavorable outcome using a composite variable strategy.
Time Frame: Baseline, Day 150
Population: Full Analysis Set, all randomized participants with a valid assessment for the outcome measure.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Ratio from baseline
Arm/Group | Inclisiran | Ezetimibe | Placebo
Number analyzed (Participants) | 173 | 88 | 87
Ratio from baseline
  LS Mean (Treatment Policy estimand) | 0.690 [0.611 to 0.780] | 0.911 [0.830 to 1.000] | 0.923 [0.803 to 1.060]
  LS Mean (Monotherapy estimand) | 0.687 [0.612 to 0.722] | 0.912 [0.836 to 0.95] | 0.922 [0.800 to 1.062]
Statistical Analysis 1: Comparison: Inclisiran vs Ezetimibe; Treatment Policy Estimand; Test type: Superiority; p = 0.0002, ANCOVA; Ratio of Geometric Mean = 0.757, 95% CI 2-sided [0.650 to 0.882]
Statistical Analysis 2: Comparison: Inclisiran vs Placebo; Treatment Policy Estimand; Test type: Superiority; p = 0.0010, ANCOVA; Ratio of Geometric Mean = 0.748, 95% CI 2-sided [0.622 to 0.898]
Statistical Analysis 3: Comparison: Inclisiran vs Ezetimibe; Monotherapy Estimand; Test type: Superiority; p < 0.0001, ANCOVA; Ratio of Geometric Mean = 0.753, 95% CI 2-sided [0.652 to 0.871]
Statistical Analysis 4: Comparison: Inclisiran vs Placebo; Monotherapy Estimand; Test type: Superiority; p = 0.0008, ANCOVA; Ratio of Geometric Mean = 0.746, 95% CI 2-sided [0.622 to 0.893]

9. Secondary Outcome: Incidence of Treatment Emergent Adverse Events (TEAE) and Serious Adverse Events (SAE)
Description: Incidence of TEAEs (regardless of seriousness) and SAEs by treatment group, including changes in laboratory results qualifying and reported as AEs.
Time Frame: From first dose of study treatment on Day 1 up to Day 180
Population: Safety Analysis Set, all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Inclisiran | Ezetimibe | Placebo
Number analyzed (Participants) | 174 | 89 | 87
Participants
  AEs | 54 | 27 | 25
  AEs related to s.c. treatment (Inclisiran or s.c. matching placebo) | 11 | 4 | 0
  AEs related to p.o. treatment (ezetimibe or p.o. matching placebo) | 3 | 2 | 2
  SAEs | 1 | 0 | 0
  SAEs related to s.c. treatment (Inclisiran or s.c. matching placebo) | 0 | 0 | 0
  SAEs related to p.o. treatment (ezetimibe or p.o. matching placebo) | 0 | 0 | 0
  Fatal SAEs | 0 | 0 | 0
  AEs leading to treatment discontinuation of inclisiran or s.c. matching placebo | 3 | 0 | 0
  AEs leading to treatment discontinuation of ezetimibe or p.o. matching placebo | 4 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study treatment on Day 1 up to Day 180
Groups:
- Total: Total
Arm/Group | Inclisiran | Ezetimibe | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/174 | 0/89 | 0/87 | 0/350
Serious Adverse Events (participants affected / at risk) | 1/174 | 0/89 | 0/87 | 1/350
Other Adverse Events (participants affected / at risk) | 19/174 | 18/89 | 13/87 | 50/350
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inclisiran (N=174) | Ezetimibe (N=89) | Placebo (N=87) | Total (N=350)
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inclisiran (N=174) | Ezetimibe (N=89) | Placebo (N=87) | Total (N=350)
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 2 | 5
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0 | 4
COVID-19 (Infections and infestations) | 1 | 2 | 3 | 6
Gastroenteritis (Infections and infestations) | 2 | 2 | 0 | 4
Nasopharyngitis (Infections and infestations) | 6 | 3 | 3 | 12
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 1 | 5
Urinary tract infection (Infections and infestations) | 3 | 2 | 2 | 7
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 3
Blood pressure increased (Investigations) | 1 | 2 | 0 | 3
Headache (Nervous system disorders) | 6 | 0 | 0 | 6
Hypertonic bladder (Renal and urinary disorders) | 0 | 2 | 0 | 2
Hypertension (Vascular disorders) | 1 | 1 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT05763875/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT05763875/SAP_001.pdf